CLINICAL TRIAL: NCT00949481
Title: Increasing Family Planning Uptake Among Postpartum Women: Testing Supply and Demand Solutions
Brief Title: Increasing Family Planning Uptake Among Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Ghana Health Services (Other Government); Ministry of Health, Zambia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10083
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Postpartum Period
Keywords: postpartum; family planning; job aid; immunization; pregnancy test
MeSH Terms: interventions — Pregnancy Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Supply (Experimental): In each country, this arm will be comprised of women attending family planning clinics within the 5 facilities randomized to this group.
  Interventions: Other: Pregnancy Test
- Demand (Experimental): In each country, this arm will be comprised of women attending immunization clinics within the 5 facilities randomized to this group.
  Interventions: Other: Job aid
- Control (No Intervention): In each country, this arm will be comprised of women attending family planning and immunization clinics in 5 facilities randomized to this group.

INTERVENTIONS:
Other: Pregnancy Test — Free pregnancy test strips will be supplied to family planning clinics
  Arms: Supply
Other: Job aid — A new job-aid will be given to immunization providers that will guide them in assessing a mother's risk for pregnancy (based on LAM criteria), and guide them in making family planning referrals, including when a woman should start to use a family planning method if she wants to prevent pregnancy. The providers in immunization clinics will be asked to make such an assessment each time a woman has her baby vaccinated.
  Additionally, in family planning clinics located in the same facilities as the immunization clinics, family planning providers will be trained to use and provided with the pregnancy checklist (see "links" for more information on the checklist)
  Arms: Demand

SUMMARY:
The rationale for the study stems from the goal of reducing the very high unmet need for family planning among women in their first year postpartum. It is understood that the reason this need is so high in general is because postpartum women do not always "demand" family planning services, and family planning providers do not always "supply" services to postpartum (amenorrheic) women who do "demand" them. To address these supply and demand problems, corresponding supply and demand solutions will be tested.

1. Demand Generating Strategy-Integrate into Immunization Services Following birth, return to fertility among postpartum women is dependent on many factors. These include time since last birth, breastfeeding intensity, and menstrual status. However, when and how fertility returns is often misunderstood by women. For instance, many women think that they can not get pregnant before their menses return, or that as long as they are breastfeeding they are protected from pregnancy. Educating women about their return to fertility following giving birth, and reminding women about the importance of birth spacing for their health and the health of their children is the focus of the demand-generating strategy.

   To reach postpartum women with these messages a demand generating activity at immunization clinics will be conducted, as immunization services are well attended. Based on the recommended immunization schedules for infants, women will make several visits to these clinics throughout the course of their first year postpartum, which provides an ideal opportunity to "hit" them with family planning messages more than once.

   To aid providers of immunization services in their delivery of family planning messages, a simple job aid was developed. The job aid takes providers through a series of 3 questions that will allow the provider to determine a mother's immediate risk for pregnancy (based on LAM criteria). If a woman is currently at risk for pregnancy, it prompts the provider to give a healthy timing and spacing message and to make a referral to the family planning clinic. If a woman is not currently at risk for pregnancy, the job aid helps the provider instruct the mother about when her risk for pregnancy will change, and therefore when she will need to seek family planning services to achieve proper birth spacing (should this be desirable to the mother).

   Also, in the family planning (FP) clinics that are located in the same facility as the immunization clinic, providers will be given the pregnancy checklist. This job-aid has already been researched (refer to citations). The purpose of providing it is to make sure that when women are referred to FP clinics by immunization providers, FP providers will supply them with a method. As a consequence, it hoped that by the time women are 9-12 months postpartum, there will be an increase in uptake of non-condom family planning methods.
2. Supply Solution-Diversify Tools Available to Rule-Out Pregnancy The supply strategy focuses on giving providers the tools to give contraceptive methods to women who are amenorrheic. As recommended by the WHO, it is standard practice for FP providers to rule out the possibility of pregnancy before providing many types of methods to their clients. The presence of menses is often used to make this determination. However, return of menses can be delayed for many months in the postpartum period, limiting a provider's ability to supply postpartum women with contraceptive methods. To overcome this challenge, the Pregnancy Checklist was developed. It is a job-aid designed to rule out pregnancy based on client responses to questions concerning her recent sexual and reproductive history. Urine pregnancy testing is another viable option for ruling out pregnancy in non-menstruating FP clients, especially in situations where providers feel they cannot trust women to answer questions honestly. Thus, family planning clinics will be provided with free pregnancy test strips, and the change in same day uptake of FP methods will be measured.

Hypotheses

1. Providing family planning messages to women attending immunization clinics with their child will cause them to seek family planning services in a greater proportion at 9-12 postpartum.
2. The availability of free pregnancy testing will increase same day method provision for new and restarting family planning clients.

ELIGIBILITY:
Inclusion Criteria:

* New and restarting family planning client (women seeking family planning service)
* Women with children 9-12 months of age attending immunization services

Exclusion Criteria:

* Attending immunization services with a child other than one's own

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14050 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The difference in current use of a modern family method among women attending immunization clinics for a child 9 to 12 months old between arms 2 and 3 of the study. | 13 months
The difference in immediate uptake of a modern family planning method (excluding condoms) among new and re-starting family planning clients between arms 1 and 3 of the study. | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Central Region, GHANA, Cape Coast, Central Region, Ghana
- Central Province, ZAMBIA, Kabwe;Chibombo, Central Province, Zambia

REFERENCES:
- [Background] Stanback J, Qureshi Z, Sekadde-Kigondu C, Gonzalez B, Nutley T. Checklist for ruling out pregnancy among family-planning clients in primary care. Lancet. 1999 Aug 14;354(9178):566. doi: 10.1016/S0140-6736(99)01578-0. PMID 10470704
- [Derived] Vance G, Janowitz B, Chen M, Boyer B, Kasonde P, Asare G, Kafulubiti B, Stanback J. Integrating family planning messages into immunization services: a cluster-randomized trial in Ghana and Zambia. Health Policy Plan. 2014 May;29(3):359-66. doi: 10.1093/heapol/czt022. Epub 2013 Apr 9. PMID 23570834